CLINICAL TRIAL: NCT02576938
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of Baricitinib in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16284; I4V-MC-JAHG (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — baricitinib; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib (Experimental): Administered once daily in multiple oral dose cohorts for 16 weeks
  (Triamcinolone 0.1% topical also permitted)
  Interventions: Drug: Baricitinib; Drug: Triamcinolone (Optional)
- Placebo (Placebo Comparator): Administered orally once daily, for 16 weeks
  (Triamcinolone 0.1% topical also permitted)
  Interventions: Drug: Placebo; Drug: Triamcinolone (Optional)

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104; INCB028050
  Arms: Baricitinib
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Triamcinolone (Optional) — Administered topically

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Baricitinib in eczema.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate-to-severe Atopic Dermatitis (AD), as determined by all of the following:

  1. EASI of 12 or more
  2. Greater than or equal to 10% of body surface area involvement
  3. Diagnosed with AD at least 2 years prior
* Have a history of inadequate clinical response to other eczema treatments

Exclusion Criteria:

* Females who are pregnant or nursing
* Participants who do not agree to use adequate contraception
* Are currently experiencing or have a history of:

  * Skin conditions such as psoriasis or lupus erythematosus
  * Skin disease that requires frequent hospitalizations or intravenous treatment
  * Compromised immunity
* Serious illness that could interfere with study participation, or a clinically important deviation in physical examination, vital sign measurements, electrocardiograms, or abnormalities on laboratory tests
* Currently experiencing or have a history of:

  * Active or latent Tuberculosis or specific immunity disorders and infections
  * Malignancy or lymphoproliferative diseases in the last 5 years (or cervical, basal or squamous skin cancer re-occurrence in the last 3 years)
  * Human Immunodeficiency Virus (HIV)
  * Hepatitis B, Hepatitis C, or chronic liver disease
* Have received certain types of vaccinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-02; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (9):
  - Dermatology Research Associates, Los Angeles, California
  - Forward Clinical Trials, Inc, Tampa, Florida
  - Medical Dermatology Specialists, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Icahn School of Medicine, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Takaoka-shi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Katoh N, Takita Y, Isaka Y, Nishikawa A, Torisu-Itakura H, Saeki H. Pooled Safety Analysis of Baricitinib in Adult Participants with Atopic Dermatitis in the Japanese Subpopulation from Six Randomized Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2765-2779. doi: 10.1007/s13555-022-00828-5. Epub 2022 Oct 18. PMID 36255569
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- See also: Click here for more information about this study: A Study of Baricitinib (LY3009104) in Participants With Moderate-to-Severe Atopic Dermatitis — http://www.lillytrialguide.com/EN-us/studies/atopic-dermatitis/jahg

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD), for 16 weeks. Triamcinolone 0.1% applied topically also permitted throughout study.
- 2 mg Baricitinib: 2 milligram (mg) Baricitinib administered PO QD for 16 weeks. Triamcinolone 0.1% applied topically also permitted throughout study.
- 4 mg Baricitinib: 4 mg Baricitinib administered PO QD for 16 weeks. Triamcinolone 0.1% applied topically also permitted throughout study.
Period: Overall Study
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Started | 49 | 37 | 38
Received at Least One Dose of Study Drug | 49 | 37 | 38
Completed | 29 | 25 | 26
Not Completed | 20 | 12 | 12
Not completed — Adverse Event | 5 | 3 | 6
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 4
Not completed — Lack of Efficacy | 9 | 4 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Met Exclusion Criteria | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD), for 16 weeks Triamcinolone 0.1% applied topically also permitted throughout study.
- 2 mg Baricitinib: 2mg Baricitinib administered PO QD for 16 weeks. Triamcinolone 0.1% applied topically also permitted throughout study.
- 4mg Baricitinib: 4mg Baricitinib administered PO QD for 16 weeks. Triamcinolone 0.1% applied topically also permitted throughout study.
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib | Total
Number analyzed (Participants) | 49 | 37 | 38 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.49) | 40.0 (14.38) | 36.4 (14.47) | 37.8 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 16 | 56
  Male | 24 | 22 | 22 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 6 | 14
  Not Hispanic or Latino | 45 | 33 | 32 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 8 | 9 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
  Black or African American | 7 | 9 | 9 | 25
  White | 23 | 20 | 18 | 61
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 31 | 32 | 105
  Japan | 8 | 6 | 6 | 20
Median EASI Total Score [Median (Full Range); unit: units on a scale] — The Eczema Area and Severity Index (EASI) assesses extent of disease based on dividing the skin into 4 regions (head/neck, trunk, upper limbs, and lower limbs) and measures the following clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3.The EASI confers a maximum score of 72 with 0 = clear; 0.1 -1 = almost clear; 1.1 -7 = mild; 7.1 - 21 = moderate; 21.1 - 50 = severe; 50.1 - 72 = very severe.
  units on a scale | 22.1 [12.0 to 70.3] | 22.1 [12.2 to 72.0] | 19.5 [12.2 to 71.4] | 21.2 [12.0 to 72.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 50% or Greater Reduction in the Eczema Area and Severity Index (EASI 50)
Description: The EASI 50, defined as ≥ 50% reduction from baseline in EASI score, assesses extent of disease based on dividing the skin into 4 regions (head/neck, trunk, upper limbs, and lower limbs) and measures the following clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3.The EASI confers a maximum score of 72 with 0 = clear; 0.1 -1 = almost clear; 1.1 -7 = mild; 7.1 - 21 = moderate; 21.1 - 50 = severe; 50.1 - 72 = very severe.
Time Frame: Week 16
Population: All participants who received at least one dose of study drug and had EASI 50 data at Week 16.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 37 | 38
percentage of participants | 37 | 57 | 61
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.065, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p = 0.027, Chi-squared

2. Secondary Outcome: Change From Baseline in the EASI at Week 16
Description: The Eczema Area and Severity Index (EASI) assesses extent of disease based on dividing the skin into 4 regions (head/neck, trunk, upper limbs, and lower limbs) and measures the following clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3.The EASI confers a maximum score of 72 with 0 = clear; 0.1 -1 = almost clear; 1.1 -7 = mild; 7.1 - 21 = moderate; 21.1 - 50 = severe; 50.1 - 72 = very severe. Change from baseline were analyzed with a Mixed-effect Model Repeated Measure (MMRM) with fixed effects for treatment, visit, country, and the treatment-by-visit interaction, plus baseline and baseline-by-visit included as covariates.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 37 | 38
units on a scale | -10.84 (1.62) | -16.44 (1.72) | -16.04 (1.72)

3. Secondary Outcome: Percentage Change From Baseline in the EASI at Week 16
Description: The Eczema Area and Severity Index (EASI) assesses extent of disease based on dividing the skin into 4 regions (head/neck, trunk, upper limbs, and lower limbs) and measures the following clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3.The EASI confers a maximum score of 72 with 0 = clear; 0.1 -1 = almost clear; 1.1 -7 = mild; 7.1 - 21 = moderate; 21.1 - 50 = severe; 50.1 - 72 = very severe. Changes from baseline were analyzed with an MMRM with fixed effects for treatment, visit, country, and the treatment-by-visit interaction, plus baseline and baseline-by-visit included as covariates.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 37 | 38
units on a scale | -45.87 (5.85) | -64.19 (6.20) | -64.69 (6.21)

4. Secondary Outcome: Change From Baseline in the Scoring Atopic Dermatitis (SCORAD) at Week 16
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates five clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation and (5) lichenification. SCORAD also assesses subjective symptoms of pruritus and sleep loss with Visual Analogue Scales (VAS) where 0 is no itch (or sleeplessness) and 10 is the worst imaginable itch (or sleeplessness). These three aspects: extent of disease (A: 0-102), disease severity (B: 0-18) and subjective symptoms (C:0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103 where 0 = no disease and 103 = severe disease. Changes from baseline were analyzed with an MMRM with fixed effects for treatment, visit, country, and the treatment-by-visit interaction, plus baseline and baseline-by-visit included as covariates.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 37 | 38
units on a scale | -11.89 (2.88) | -23.87 (3.03) | -26.54 (2.97)

5. Secondary Outcome: Change From Baseline in the Investigator's Global Assessment (IGA) at Week 16
Description: The IGA consists of a 6-point severity scale to measure characteristics of erythema, infiltration, papulation, oozing and crusting as guidelines for the overall severity assessment. The scale ranges from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease and 5 = very severe disease).
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug and had IGA data at Week 16 .
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 29 | 27 | 29
units on a scale | -0.9 (0.69) | -1.4 (1.31) | -1.3 (1.01)

6. Secondary Outcome: Change From Baseline in the Dermatologic Life Quality Index (DLQI) at Week 16
Description: The DLQI is a simple, participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". For all questions, if unanswered the question is scored as "0". Totals range from 0 to 30 (less to more impairment). Changes from baseline in DLQI score were analyzed with an MMRM with fixed effects for treatment, time, country, and the treatment-by-visit interaction, plus baseline and baseline-by-visit were included as covariates.
Time Frame: Baseline, Week 16
Population: All participants who have received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 37 | 38
units on a scale | -6.27 (0.82) | -6.89 (0.89) | -7.96 (0.86)

7. Secondary Outcome: Change From Baseline in the Itch Numerical Rating Scale (NRS) at Week 16
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by circling the number that best describes the worst level of itching in the past 24 hours. Changes from baseline were analyzed with an MMRM with fixed effects for treatment, time, country, and the treatment-by-visit interaction, plus baseline and baseline-by-visit were included as covariates.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 37 | 38
units on a scale | -1.72 (0.44) | -2.61 (0.47) | -2.22 (0.46)

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Baricitinib
Description: Pharmacokinetics (PK): Maximum serum concentration (Cmax) of Baricitinib
Time Frame: Week (Wk) 0: Predose, 15-30 minutes (min) postdose; Wk 4: 1.5 - 4 hour (hr) postdose; Wk 8: 4 - 8 hr postdose; Wk 12: Predose; Wk 16: 30 - 90 min postdose.
Population: All participants who received at least 1 dose of study drug and provided at least 1 post-dose PK sample. PK sample was not collected for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 2 mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 37 | 38
nanogram per milliliter (ng/mL) | 18.5 (70.0) | 37.7 (38.9)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 5 months)
Arm/Group | Placebo | 2 mg Baricitinib | 4mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/49 | 2/37 | 1/38
Other Adverse Events (participants affected / at risk) | 14/49 | 13/37 | 19/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | 2 mg Baricitinib (N=37) | 4mg Baricitinib (N=38)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | 2 mg Baricitinib (N=37) | 4mg Baricitinib (N=38)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 3 (4) | 1 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 5 (5)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 5 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (6):
  • Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT02576938/SAP_000.pdf
  • Study Protocol: Protocol (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT02576938/Prot_001.pdf
  • Study Protocol: Protocol Amendment (a) (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02576938/Prot_002.pdf
  • Study Protocol: Protocol Amendment (b) (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT02576938/Prot_003.pdf
  • Study Protocol: Protocol Amendment (c) (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02576938/Prot_004.pdf
  • Study Protocol: Protocol Amendment (d) (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT02576938/Prot_005.pdf